CLINICAL TRIAL: NCT02863367
Title: A One-Arm Exploratory Clinical Trial of Apatinib Plus Gemcitabine in Patients With Advanced Metastatic Pancreatic Cancer
Acronym: OECTAPGAMPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBP001
Record Dates: First submitted 2016-07-26; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — apatinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Apatinib：500 mg，po，qd, d1-14, every 3 week Gemcitabine：1000mg/m²，vein input 30-40，d1，d8，every 3 week
  Interventions: Drug: Apatinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Apatinib — Apatinib：500 mg，po，qd, d1-14, every 3 week
  Other Names: YN968D1
Drug: Gemcitabine — Gemcitabine：1000mg/m²，vein input 30-40，d1，d8，every 3 week

SUMMARY:
Evaluate the efficacy and safety of Apatinib (500mg/d) with gemcitabine(1000mg/m2) in advanced metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This test is a single center, one-armed exploratory clinical research, aimed at the evaluation the efficacy and safety of Apatinib with Gemcitabine in the patients with advanced metastatic pancreatic cancer.

This study plan in Tianjin Medical University Cancer Institute and Hospital.From launched in July 2016, this research intends to recruit the end time about as of December 2017, is expected to the end of the test time is in December 2017.

If do not have the appearance of the following circumstances, such as the subjects out of informed consent, drug toxicity tolerance or the researchers think that do not fit for further test, each subject research and treatment time is expected until imaging of tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients ranges from 18 to 75 years old.
2. Histologically or cytologic confirmed advanced metastatic pancreatic cancer (Exclusion of islet cell tumor ) .
3. Must not received radiotherapy, chemotherapy or experimental treatment for advanced metastatic pancreatic cancer. Transfer of postoperative recurrence of patients with advanced pancreatic cancer can also be into the group.
4. Karnofsky Performance Status Scale (KPS) ≥70.
5. The first confirmed date of advanced metastatic pancreatic cancer not more than 6 weeks before starting treatment.
6. No jaundice symptoms. Obviously abdominal water or have symptoms, need a drainage in advance. Don't need to adjust the analgesic therapy.
7. Adequate hematologic functions :Hemoglobin (HGB) ≥ 90g/dL, Platelets (PLT) ≥ 100×10^9/L, the absolute number of Neutrophil (ANC) ≥ 1.5×10^9/L.
8. Adequate hepatic, renal, heart functions :Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×the upper limit of normal (ULN).If liver metastases, AST and ALT ≤5.0×the ULN. Total bilirubin within the ULN. Serum Creatinine within the ULN, or creatinine clearance ≥ 60 mL/min.
9. Blood coagulation test results: Prothrombin Time (PT) and Partial Thromboplastin Time (PPT) within ±15% of the normal.
10. No clinically significant abnormal urine analysis results.
11. Women with pregnancy or lactation, or fertility but during treatment and 6 months after treatment of termination unwilling or unable to use effective contraception to avoid pregnancy patients with male or female
12. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
13. Patient consent and well compliance, scheduled to accept the visits, treatment, laboratory tests and other study procedures

Exclusion Criteria:

1. Patients with the known brain metastases.
2. Patients with locally advanced disease only.
3. Decline in serum albumin (ALB) ≥ 20% from the screening visit to cycle 1 day 1 prior to the 72 hours.
4. Over the past five years has a history of malignant tumors (including chronic leukemia). Patients with carcinoma in situ or basal cell carcinoma or squamous cell skin cancer can be selected.
5. With need of systemic treatment activity, unable to control bacterial, viral or fungal infections
6. Known HIV infection, or active hepatitis B or hepatitis C virus (HCV) infection.
7. A major surgery (not include the diagnostic surgery) not more than 4 weeks before starting treatment.
8. In the period of 6 months before starting treatment, Patients with myocardial infarction, severe or unstable angina, coronary artery and peripheral artery bypass grafting, New York heart association (NYHA) three - four level cardiac failure, out of control of high blood pressure, Patients with clinical significance of arrhythmia or abnormal electrocardiogram (ECG), cerebrovascular accident, transient ischemic attack, epilepsy, or with clinical significance of arrhythmia or a history of abnormal electrocardiogram (ECG).
9. Has any study drug or its accessories history of allergies or allergic reactions, or patients showed this product or controlled drug prescribing information "contraindications or special warnings and precautions" section Outlines of events.
10. The history of connective tissue disease (such as lupus, scleroderma, nodular arteritis).
11. Has a history of interstitial pneumonia, slowly progressive dyspnea and cough, sarcoidosis, and silicosis, idiopathic pulmonary fibrosis, hypersensitivity pneumonitis, or a variety of allergies.
12. Could damage patient safety or the integrity of the data to any situation, including severe medical risk factors, medical events and laboratory abnormalities or mental illness;
13. Enter any other clinical study, some involved in drug test, or may interfere with the study in the program evaluation;
14. The patient is not willing to or cannot meet research program, or plans for vacation during the research and treatment more than 7 days or seven days;
15. The investigator think that the person doesn't fit into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 years

SECONDARY OUTCOMES:
progression-free survival (PFS) | 1 years
Overall Survival (OS) | 1 years
Life Quality Score (QoL) | 1 years
Disease Control Rate (DCR) | 1 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Hao Ji Hui, PhD, Principal Investigator — National Clinical Research Center for Cancer of China

IPD SHARING:
Plan to Share IPD: Undecided